CLINICAL TRIAL: NCT02746562
Title: A Multicentre Randomized Controlled Trial of a "Freeze All and Transfer Later" Versus a Conventional "Fresh Embryo Transfer" Strategy for Assisted Reproductive Technology (ART) in Women With a Regular Menstrual Cycle
Brief Title: Study Comparing Outcomes Between Conventional IVF and a "Freeze-all"-Strategy in Assisted Reproductive Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anja Bisgaard Pinborg (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other); Holbaek Sygehus (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other); Regional Hospital Skive (Unknown); Dexeus University Hospital Barcelona (Unknown)
Responsible Party: Sponsor-Investigator, Anja Bisgaard Pinborg, Professor, MD, DMSc, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1600-1116
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Infertility
Keywords: Assisted reproduction; In vitro fertilisation; Frozen embryo transfer (FET)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freeze all (Experimental): Transfer of a frozen, thawed blastocyst in a subsequent natural menstrual cycle
  Interventions: Procedure: Freeze all
- Fresh embryo transfer (No Intervention): Standard procedure

INTERVENTIONS:
Procedure: Freeze all — Freezing of all blastocyst stage embryos with thawing and transfer in a subsequent natural cycle
  Arms: Freeze all

SUMMARY:
The purpose of this study is to compare conventional fresh embryo transfer with a "freeze all and transfer later strategy" in assisted reproductive technology in terms of ongoing pregnancy rates, live birth rates as well as perinatal outcomes.

DETAILED DESCRIPTION:
The study is a multicentre randomized controlled double-blinded trial with the purpose to investigate if pregnancy- and live birth rates can be improved by a "freeze all and transfer later"-strategy with transfer of the best quality, frozen, thawed embryo in a subsequent natural cycle compared with conventional fresh embryo transfer with transfer of the embryo in the stimulated cycle.

In total 5 clinics in Denmark and Sweden will be participating in the recruitment of patients for the study.

The patients will be screened and randomized computerized on cycle day 2 or 3 and allocated to one of the two study arms:

I: hCG (human chorion gonadotrophin) arm with traditional hCG triggering and fresh blastocyst transfer II: GnRH (gonadotropin-releasing hormone)- agonist triggering arm with blastocyst cryopreservation and subsequent transfer in a subsequent natural cycle.

The randomization will be done after the decision of gonadotrophin (rFSH/hMG) starting dose, and both doctor and patient will be blinded to the randomization until the day of hCG/agonist trigger. Both groups will be stimulated in a short GnRH antagonist protocol. The ovarian stimulation The gonadotrophin stimulation is performed according to the general standards in each of the clinics and can be altered according to the ovarian response with a maximum of 300 IU.

Blood samples are collected at baseline before the first gonadotrophin injection and at day of hCG injection and further blood samples in the luteal phase will be collected for a small subgroup of patients. All blood samples will be kept at the Biobank for the study at Hvidovre Hospital.

Women in both arms will furthermore be requested to fill out a physical discomfort and a quality of life questionnaire at two different visits. Additionally the men will be asked to fill out quality of life questionnaires.

Comprehensive sonography will be performed at the start of ovulation with details on each ovary. Ultrasound examination is performed on cycle day 2-3, at stimulation day 6 and thereafter every 2-3 days until ovulation is inducted.

On the day of oocyte retrieval the randomization is unblinded. The oocytes are fertilized by either IVF or ICSI and cultured individually according to the normal procedures in the clinics.

If the patient is allocated to the "Fresh embryo transfer"-group the best quality blastocyst will be transferred on day five after oocyte pick-up, if a blastocyst is developed. Surplus good quality blastocysts are vitrified on day five or six.

For patients in the "Freeze all" group all embryos of good quality are vitrified at the blastocyst stage day 5 in the stimulated cycle according to the criteria for freezing blastocysts in each clinic. The highest quality embryo is selected and marked and will be the first one to be thawed after at least one mentrual cycle that is considered as a wash out period. Embryo transfer is performed 6-7 days after hCG injection in the blastocyst transfer cycle in this group.

A serum beta-hCG test is performed 11 days after blastocyst transfer, and clinical pregnancy is confirmed by transvaginal ultrasound 3 to 4 weeks after a positive serum-hCG test.

A follow-up of all pregnancies will be performed within three months after delivery or termination of pregnancy on predefined information sheets. All pregnancies resulting from blastocysts retrieved and thawed according to this study protocol will be followed from study inclusion and one year onwards.

All data will be collected in a single database and all participants will be anonymized by way of an identificationcode. The biobank will be closed and all samples destroyed after 5 years of the conclusion of the study at the latest.

The study is a superiority study with 424 (212 in each arm) patients required to have an 80 % chance of detecting, as significant at the 5 % level, a decrease in the primary outcome measure from 30 % in the control group to 43 % in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* AMH (Anti-Müllerian hormone) > 6.28 pmol/L (Roche Elecsys assay)
* Female age 18 years to less than 40 years
* 1, 2 or 3 IVF/ICSI cycle with oocyte aspiration
* Regular menstrual cycle between 24 and 35 days
* BMI between 18 and 35
* Two ovaries
* Can and will sign informed consent

Exclusion Criteria:

* Women who do not fulfil the inclusion criteria
* Endometriosis stage III to IV
* Ovarian cysts with diameter > 30 mm at day of start of stimulation
* Submucosal fibroids
* Women with severe co-morbidity (IDDM, NIDDM, gastrointestinal, cardiovascular, pulmonary, liver or kidney disease)
* Dysregulation of thyroid disease
* Not danish or English speaking women
* Contraindications or allergies to use of Gonadotrophins or GnRH antagonists
* TESA (testicular sperm aspiration)
* OD (oocyte donation)
* Previous inclusion in the study

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 424 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | Two years
  Outcome measured per transfer of the first blastocyst, per oocyte pick-up, per start of ovarian stimulation and per randomized patient.

SECONDARY OUTCOMES:
Live birth rates | Two years
  Outcome measured after the first blastocyst transfer calculated per randomized patient, per started ovarian stimulation, per oocyte pick-up and per transfer
Cumulative live birth rates | Two years
  Measured after one stimulated cycle with oocyte retrieval and after use of all frozen blastocysts or after at least 1 year of follow-up
Number of cycles with no embryo transfer | Two years
Time-to-pregnancy | Two years
  From start of ovarian stimulation to positive hCG
Time-to-delivery | Three years
Preterm birth | Three years
Low birth weight | Three years
Small-for-gestational age (SGA) | Three years
Large-for-gestational age (LGA) | Three years
Perinatal mortality | Three years
Preeclampsia | Three years
Placental rupture | Three years
Positive hCG 11 days post embryo transfer | Three years
Miscarriages, biochemical pregnancies, ectopic pregnancies | Three years
Quality of life for female and partner | Two years
Cost-effectiveness | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bisgaard Pinborg, MD, DMSc, Study Director — Fertility Clinic, Obstetrical and Gynecological department, Hvidovre Hospital
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - University Hospital Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilegaard SP, Schmidt L, Stormlund S, Koert E, Bogstad JW, Praetorius L, Nielsen HS, la Cour Freiesleben N, Sopa N, Klajnbard A, Humaidan P, Bergh C, Englund ALM, Lossl K, Pinborg A. Psychosocial wellbeing shortly after allocation to a freeze-all strategy compared with a fresh transfer strategy in women and men: a sub-study of a randomized controlled trial. Hum Reprod. 2023 Nov 2;38(11):2175-2186. doi: 10.1093/humrep/dead188. PMID 37742131
- [Derived] Alexopoulou E, Stormlund S, Lossl K, Praetorius L, Sopa N, Bogstad JW, Mikkelsen AL, Forman J, la Cour Freiesleben N, Vikkelso Jeppesen J, Bergh C, Al Humaidan PSH, Grondahl ML, Zedeler A, Pinborg AB. Embryo Morphokinetics and Blastocyst Development After GnRH Agonist versus hCG Triggering in Normo-ovulatory Women: a Secondary Analysis of a Multicenter Randomized Controlled Trial. Reprod Sci. 2021 Oct;28(10):2972-2981. doi: 10.1007/s43032-021-00564-9. Epub 2021 Apr 13. PMID 33847977
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Stormlund S, Sopa N, Zedeler A, Bogstad J, Praetorius L, Nielsen HS, Kitlinski ML, Skouby SO, Mikkelsen AL, Spangmose AL, Jeppesen JV, Khatibi A, la Cour Freiesleben N, Ziebe S, Polyzos NP, Bergh C, Humaidan P, Andersen AN, Lossl K, Pinborg A. Freeze-all versus fresh blastocyst transfer strategy during in vitro fertilisation in women with regular menstrual cycles: multicentre randomised controlled trial. BMJ. 2020 Aug 5;370:m2519. doi: 10.1136/bmj.m2519. PMID 32759285
- [Derived] Stormlund S, Lossl K, Zedeler A, Bogstad J, Praetorius L, Nielsen HS, Bungum M, Skouby SO, Mikkelsen AL, Andersen AN, Bergh C, Humaidan P, Pinborg A. Comparison of a 'freeze-all' strategy including GnRH agonist trigger versus a 'fresh transfer' strategy including hCG trigger in assisted reproductive technology (ART): a study protocol for a randomised controlled trial. BMJ Open. 2017 Jul 31;7(7):e016106. doi: 10.1136/bmjopen-2017-016106. PMID 28760794